CLINICAL TRIAL: NCT05730348
Title: Mealtime Anxiety in Eating Disorders: An Ecological Momentary Assessment (EMA) Project
Brief Title: Mealtime Anxiety in Eating Disorders
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Dam Foundation (Other)
Responsible Party: Principal Investigator, Kristin Stedal, Researcher, Oslo University Hospital
Other Study IDs: 541774
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with eating disorders
  Interventions: Behavioral: Post mealtime activity

INTERVENTIONS:
Behavioral: Post mealtime activity — Therapist lead movement post meals

SUMMARY:
The goal of this observational study is to assess mealtime anxiety in patients with eating disorders receiving treatment at an in-patient unit. Anxiety wil be assessed using ecological momentary assessment (EMA). The main research question is:

• Does post meal activity reduce anxiety in patients with eating disorders?

Study participation will last for two weeks. Participants will be reporting current levels of anxiety/distress on an EMA mobile app during treatment as usual. During one of the two study participation weeks, the participants will perform post mealtime activity.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Regional Department for Eating Disorders adult in-patient unit (>16 years old) will be invited to participate.

Exclusion Criteria:

* Patients who receive tube feeding for all meals during the study period will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be patients suffering from eating disorders, treated at a specialized eating disorder unit, at tertiary level of health care. The population is expected to primarily consist of individuals suffering from anorexia nervosa, but all patients admitted to the ward will be invited to participate, independent of eating disorder diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Self Reported Anxiety During Treatment as Usual vs Treatment as Usual plus Post-Mealtime Activity | Two weeks
  Anxiety will be measured using the Subjective Units of Distress Scale (SUDS). Higher scores indicate higher levels of distress. The Affect Grid will also be used to assess current mood. Measures will be collected using Ecological Momentary Assessment (EMA).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Stedal, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Regional Department for Eating Disorders, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No